CLINICAL TRIAL: NCT04684823
Title: The Impact of Patch Rx Technologies on Adherence to Vitamin and Trikafta® (Elexacaftor/Tezacaftor/Ivacaftor) Therapies in Patients With Cystic Fibrosis
Brief Title: The Impact of Patch Rx Technologies on Adherence to Vitamin and Trikafta Therapies in Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Patch Rx Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HSC20200875H
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Cystic Fibrosis; Adherence, Medication
MeSH Terms: conditions — Cystic Fibrosis; Medication Adherence

STUDY DESIGN:
Intervention Model Description: Single arm device pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Use of Patch Cap and Patch App (Experimental): Subjects will use Patch Technologies to track their medication regimen compliance
  Interventions: Device: Patch Cap; Device: Patch App

INTERVENTIONS:
Device: Patch Cap — A prescription container cap to track the dispensing of an oral dose of medication with an associated app which tracks the adherence to medication regimen.
Device: Patch App — A mobile app that is used with Patch Cap to track adherence to medication regimen

SUMMARY:
This proposed pilot study will assess if the Patch Technology system will increase adherence in patients with cystic fibrosis followed at the UTHSCSA Cystic Fibrosis Center.

DETAILED DESCRIPTION:
This trial will follow patients' adherence with their current medication regimen and will not impact the medications they are prescribed. Patients will be enrolled during a regularly scheduled Cystic Fibrosis Clinic visit. When participants receive their reminder calls for the clinic visit, they will be asked to bring their prescribed vitamins in the pharmacy dispensed bottle with them. During the clinic visit, the study will be reviewed, and consent will be obtained. After enrollment, patients will complete a survey indicating their understanding of the reason for taking vitamins/genetic modulators, the importance they place on taking the medications, self-reported adherence to the therapies, and reasons for being non-adherent. Participants will indicate which pharmacies they receive the vitamins and modulators from, and how they obtain the refills (E.g., Does the patient call for refills? Does the pharmacy send a reminder text/email/phone call or are medications auto refilled?) During the first visit, directions on how to download the Patch App and scan the QRS code will be sent to the subject/parent. Subjects/parents will enter their recommended dose of Trikafta and vitamin in the Patch App. Patients will be taught how to place the Patch Cap in the lid of their vitamin bottle. They will be given the option of entering data for a "buddy" who will also get a reminder when they are due to take their medications if medications are not documented as taken in a specified time window. Data which will be collected at baseline are age (< 18 years of age, > 18 years of age), gender, insurance status, Education level (parent education level if patient < 18 years of age), marital status if patient > 18 years of age, weight/BMI/FEV1 at enrollment, concomitant medications, and vitamin A and E levels measured within the previous year. Once the patient is enrolled, the study team will contact the pharmacies from which the patient gets the vitamins and elexacaftor/tezacaftor/ivacaftor and will review the refill history over the past 6 months. The study staff will calculate the Medication Possession Ration (MPR) equal to the number of pills the patient would have based on their refill history/number of pills needed to take medication as prescribed. Over the next 3 months, patients will take their medications and this activity will either be logged via the Patch Cap electronically to the Patch App or the patient will enter the data every time they take the elexacaftor/tezacaftor/ivacaftor on the Patch App. This information will simultaneously be tracked in the Patch Hub by Patch Technologies personnel. At the end of three months, patients will return to clinic for their routine quarterly visit. Patients will be surveyed about ease of use of the Patch Cap and the PatchRx App, as well as estimating their adherence. The study team will obtain the refill history for vitamins and elexacaftor/tezacaftor/ivacaftor for the previous 3 months as reported by the pharmacy and calculate the MPR. Patch Technologies will provide adherence data collected through the Patch App to the PI at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with CF and cared for at University of Texas Health San Antonio Cystic Fibrosis clinic
2. > 12 years of age
3. Prescribed a daily CF specific vitamin for at least 6 month
4. Prescribed the genetic modulator elexacaftor/tezacaftor/ivacaftor for at least 6 month
5. English speaking
6. Patient possesses a Bluetooth enabled smartphone or mobile device.

Exclusion Criteria:

1) Patient is already using some other medication therapy management (MTM) service.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Adherence to Trikafta dosing | Baseline to 90 days
  Tracking of medication compliance over the time where the Patch Cap and Patch App are used by determining number of days compliance
Adherence to Multivitamin dosing | Baseline to 90 days
  Tracking of medication compliance over the time where the Patch Cap and Patch App are used by determining number of days compliance

SECONDARY OUTCOMES:
Patch vs Self Reported Adherence for Trikafta | Baseline to 90 days
  Difference between patch cap and app measurement vs self reported adherence
Patch vs Self Reported Adherence for Multivitamin | Baseline to 90 days
  Difference between patch cap and app measurement vs self reported adherence
Median Dosing Interval | Baseline to 90 days
  Difference between median dosing interval for Trikafta using Patch App vs manufacturer recommended interval

CONTACTS AND LOCATIONS:
Overall Officials: Donna Beth J Willey-Courand, MD, Principal Investigator — UT Health San Antonio; Sarah J Kubes, Pharm D, Principal Investigator — UT Health San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States